CLINICAL TRIAL: NCT01715688
Title: Efficacy of Endotracheal Tube Cuffs Pre-filled With Alkalinized Lidocaine Compared to Endotracheal Tube Cuffs Filled With Saline on the Incidence of Coughing During Emergence of Anesthesia.
Brief Title: Efficacy of Alkalinized Lidocaine in the Endotracheal Tube Cuff on the Incidence of Coughing During Emergence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NM2012-003
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Cough; Anesthesia
MeSH Terms: conditions — Cough | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alkalinized lidocaine (Active Comparator): The endotracheal tube cuff will be pre-filled at least 90 minutes before intubation with alkalinized lidocaine. Endotracheal tube cuff will be emptied before intubation and then re-filled with the same mixture following intubation to secure the position of the endotracheal tube. (cuff will be inflated until there is no air leak around the tube).
  During emergence, when the expired fraction of desflurane reaches 0.2 MAC, the patient will be asked to open his eyes every 30 seconds. Any coughing effort before 0.2 MAC will be considered as a treatment failure and the patient will be treated according to the attending anaesthesiologist.
  Interventions: Drug: Alkalinized lidocaine
- Saline (Placebo Comparator): The endotracheal tube cuff will be pre-filled at least 90 minutes before intubation with saline. Endotracheal tube cuff will be emptied before intubation and then re-filled with the same mixture following intubation to secure the position of the endotracheal tube. (cuff will be inflated until there is no air leak around the tube).
  During emergence, when the expired fraction of desflurane reaches 0.2 MAC, the patient will be asked to open his eyes every 30 seconds. Any coughing effort before 0.2 MAC will be considered as a treatment failure and the patient will be treated according to the attending anaesthesiologist.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Alkalinized lidocaine — Administration of alkalinized lidocaine in the endotracheal tube cuff
  Arms: Alkalinized lidocaine
Drug: Saline — Administration of saline in the endotracheal tube cuff
  Arms: Saline

SUMMARY:
This study is designed to compare the efficacy of endotracheal tube cuffs pre-filled with alkalinized lidocaine on the:

* incidence of coughing during emergence of general anesthesia
* time needed for emergence following a desflurane-based anesthesia
* incidence of sore throat after extubation.

The investigator's hypothesis is that the use of endotracheal tube cuffs pre-filled with alkalinized lidocaine will reduce the incidence of coughing by 50% relative to a control group following a desflurane-based anesthesia.

DETAILED DESCRIPTION:
Emergence is an important period of general anesthesia during which several problems can occur. Coughing, hypertension, tachycardia and agitation have been observed during emergence of general anesthesia.

Desflurane is a newer volatile agent allowing early recovery from anesthesia. This agent has led to earlier discharge and more rapid resumption of normal activities after surgery. However, an incidence of coughing around 70% has been reported after a desflurane-based anesthesia. Different techniques and drugs have been studied to reduce coughing during emergence.

Among others, the role of lidocaine given intravenously, topically, or intracuff has been studied. Intracuff lidocaine has been shown to increase the tolerance to the endotracheal tube without reducing the swallowing reflex. However, lidocaine slowly diffuses across the tube's cuff. The addition of bicarbonates is required to increase its diffusion to the underlying tracheal tissue. Alkalinization of lidocaine allows the diffusion of 65% of its neutral base form over a period of 6 hours.

In vitro studies have demonstrated that the optimal time for local anesthetic diffusion through the cuff may vary from 90 to 180 minutes. Due to its low onset, this technique would be appropriate for long-duration surgeries. Pre-filling the endotracheal tube cuffs with alkalinized lidocaine at least 90 minutes before intubation could be appropriate for surgeries expected to last less than two hours.

This study will assess the efficacy of pre-filling endotracheal tube cuffs with alkalinized lidocaine to prevent coughing during emergence in short-duration surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective short-duration surgery under general anesthesia (expected duration of less than 2 hours)
* Physical status 1-3

Exclusion Criteria:

* Asthma or severe pulmonary disease
* Pulmonary tract infection
* Anticipated difficult intubation
* Current use of cough medicine
* Contraindication to lidocaine
* Pregnancy
* Airway surgery
* Inability to provide informed consent
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of coughing during emergence of general anesthesia | At extubation (Day 0)

SECONDARY OUTCOMES:
Time to emergence | At extubation (Day 0)
Incidence of sore throat | One hour after extubation (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Massicotte, MD, FRCPC, Principal Investigator — Centre Hospitalier de l'Université de Monrtréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Nath P, Williams S, Herrera Mendez LF, Massicotte N, Girard F, Ruel M. Alkalinized Lidocaine Preloaded Endotracheal Tube Cuffs Reduce Emergence Cough After Brief Surgery: A Prospective Randomized Trial. Anesth Analg. 2018 Feb;126(2):615-620. doi: 10.1213/ANE.0000000000002647. PMID 29189279